CLINICAL TRIAL: NCT06442865
Title: Freeze-dried Amniotic Membrane in the Treatment of Non-healing Wounds: a Single-arm, Retrospectivelyprospective Clinical Trial
Brief Title: AMNIODERM+ Medical Device Clinical Study
Acronym: AMNIODERM+
Status: Completed | Type: Observational
Sponsor: BioHealing s.r.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: AD+29082022ZP
Record Dates: First submitted 2024-05-23; First posted 2024-06-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Non-healing Wound; Diabetic Foot
Keywords: medical device; AMNIODERM+; non-healing wounds; DFU
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective data: Subjects with a diabetic neuropathic or neuroischemic wounds, anywhere on the leg, ranging in size between 2 cm2 and 16 cm2, that has not healed at least 20% after the 6 weeks of the standard of care (SoC) with the known therapeutic history ≥ 6 weeks and ≤ 104 weeks prior to clinical trial inclusion.
  Retrospective data will contain information about the subject's history and wound treatment by SoC.
  Interventions: Device: AMNIODERM+
- Prospective data: Subjects with a diabetic neuropathic or neuroischemic wounds, anywhere on the leg, ranging in size between 2 cm2 and 16 cm2, that has not healed at least 20% after the 6 weeks of the standard of care (SoC) with the known therapeutic history ≥ 6 weeks and ≤ 104 weeks prior to clinical trial inclusion.
  Prospective data will contain information about wound treatment by AMNIODERM+®.
  Interventions: Device: AMNIODERM+

INTERVENTIONS:
Device: AMNIODERM+ — A common surgical approach in chronic wound treatment aims at the promotion of epithelization by a combination of debridement manipulations (removal of non-vital tissues) and infection/inflammation management using antibacterial wound dressings (antibiotics or silver covering). The advantages of biomaterials can be attributed to their unique mechanical, immunological, and regenerative properties.
  The product will be evaluated in the subjects not responding to SoC.

SUMMARY:
This is retrospectively-prospective clinical trial with medical device AMNIODERM+ intended for the non-healing wounds. Retrospective data will contain information about the subject's history and wound treatment by SoC. Prospective data will contain information about wound treatment by AMNIODERM+®.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females over 18 years of age
2. Type 1 or Type 2 diabetes mellitus
3. Presence of a diabetic neuropathic or neuroischemic wound, anywhere on the leg, that has not healed at least 20% after the 6 weeks of the standard of care (SoC)
4. History of an evaluable defect ≥ 6 weeks and ≤ 104 weeks prior to clinical trial inclusion
5. Size of a wound to be evaluated 2 to 16 cm2
6. Wound treatment can be provided either on an inpatient or outpatient basis, based on the doctor's decision
7. The subject agrees to periodic visits to the clinical trial site during their participation in the clinical trial
8. The subject is able to understand the clinical trial information
9. Signed informed consent form
10. Data on previous wound care are available in the subject medical documentation

Exclusion Criteria:

1. Necrotic wound requiring surgical treatment
2. Pregnancy or breastfeeding
3. Venous etiology of ulceration
4. Burns or chemical burns
5. Clinical manifestations of systemic infection
6. Undermined wound edges
7. The wound involves deeper structures (bone, tendons, joints)
8. Inadequately controlled diabetes mellitus with HbA1c > 12 % (DCCT) diabetes mellitus
9. Renal insufficiency with eGF < 30ml/min/1.73m2
10. Infected ulceration either Stage ≥2 according to EWMA Position Document (2006) (Appendix II) or with CRP >10
11. Topical treatment with any growth factor-based products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diabetic neuropathic or neuroischemic wounds, anywhere on the leg, ranging in size between 2 cm2 and 16 cm2, that has not healed at least 20% after the 6 weeks of the standard of care (SoC) with the known therapeutic history ≥ 6 weeks and ≤ 104 weeks prior to clinical trial inclusion.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Non-healing wounds measuring | 6 + 12 weeks
  Analyses of primary and secondary endpoints: The error rate During data collection, a change was made to the CIP regarding complete wound closure (wound heal). Whether a wound was healed was determined by the opinion of the investigator and not by the size of the wound as measured by Imito® application. The error rate of the Imito® measuring application in determining the size of the wound was 10 %, i.e. based on that and clinical experience the threshold of 0.1 cm2 was determined. Wounds smaller than or equal to 0.1 cm2 were considered as complete closure. The investigator confirmed the wound closure in an accompanying comment in the eCRF.

CONTACTS AND LOCATIONS:
Locations (1):
- Národní Endokrinologický a Diabetologický ústav, Ľubochňa, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided